CLINICAL TRIAL: NCT02148029
Title: Role of a Novel Exercise Program to Prevent Post-thrombotic Syndrome
Acronym: EFFORT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0995-R
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Acute Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Post thrombotic syndrome; Thrombus resolution
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Exercise; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Standard care: anticoagulation, compression, and ad-lib ambulation
  Interventions: Other: Standard Care
- Exercise (Experimental): Standard care + Interventional Exercise therapy
  Interventions: Other: Exercise; Other: Standard Care

INTERVENTIONS:
Other: Exercise — Upper and Lower extremity exercise
  Arms: Exercise
Other: Standard Care — anticoagulation, compression, and ad-lib ambulation

SUMMARY:
Despite standard care, 25%-50% of patients with clots in the deep veins of the arms and legs progress to chronic post-clot problems resulting in significant disability, loss of productivity, and healthcare costs. Reverse flow in the veins from an organizing clot is the primary cause of post-clot problems. Veins with early clot breakdown have a lower incidence of reverse flow. The investigators have observed that clot breakdown is enhanced by increased blood flow and that moderate arm and leg exercise result in increased venous blood flow. Hence, the investigators predict that a supervised exercise program in patients with deep vein clots could increase leg vein blood flow, accelerate clot breakdown, and decrease the risk of post clot problems. The primary hypothesis is that increased blood flow across the clot (induced by supervised exercise) will increase clot breakdown and decrease severity of post clot problems. The investigators are conducting a randomized clinical trial of standard therapy compared to progressive exercise training in patients with leg deep vein clots.

DETAILED DESCRIPTION:
Standard anticoagulation therapy for acute deep vein thrombosis (DVT) reflects the current short term focus on preventing pulmonary embolism (PE) and recurrent DVT. Despite standard care, 25% to 50% of patients with DVT progress to the chronic post-thrombotic syndrome (PTS) resulting in significant disability, loss of productivity, and healthcare costs. The investigators postulate that a supervised exercise program in patients with acute DVT could increase lower extremity venous flow, accelerate thrombus resolution, and thereby decrease the risk of PTS. If the patient is unable to perform exercises, neuromuscular electrical stimulation (NMES) will be used to induce contraction of the muscles of the lower extremities.

Aim 1 will test whether a 3-month exercise program has long-term clinical benefits in acute DVT. The primary outcome measures will be the 2-year change in Villalta score for PTS and VEINES-QOL score (Venous Insufficiency Epidemiological and Economic Study-QOL).

Aim 2 will evaluate whether exercise therapy in patients with acute DVT enhances thrombus resolution. The outcome measure will be 3-month change in thrombus volume.

Aim 3 will assess the relationship between PTS, venous hemodynamics and exercise capacity. The outcome measures will be Villalta score, common femoral reflux, and 400-meter walk time.

ELIGIBILITY:
Inclusion Criteria:

* Acute Lower Extremity DVT
* DVT documented by ultrasound, CT/Magnetic Resonance imaging (MR) venogram, or conventional venogram
* Enrolled within 4 weeks of onset of symptoms
* Age 18 years or older

Exclusion Criteria:

* Peripheral arterial disease (disabling claudication, rest pain, tissue loss) with ankle brachial index (ABI)<0.5
* Immediate need for thrombolysis/thrombectomy
* DVT involving the inferior vena cava (IVC)
* Contraindication to anticoagulation
* Contraindications to exercise training
* Medical illness interfering with evaluation/follow-up
* Life expectancy <2 years
* Pregnancy
* Inability to walk
* Hemodynamically significant PE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brajesh K Lal, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (18+) patients who recently experienced acute lower extremity Deep Vein Thrombosis (DVT) were screened and enrolled within 28 days of the DVT diagnosis, received a 3-month treatment (either standard care alone or standard care + exercise program), followed for 2 years, and evaluated at 1 month, 3 months, 6 months, 1 year, and 2 years. Participants were recruited from a vascular imaging lab based on physician referral. Participants were enrolled September 2014 - June 2019.
Pre-assignment Details: Of 107 enrolled participants, 102 were randomized to one of the treatment groups.
Groups:
- Control: Standard care (anticoagulation, compression, and ad-lib ambulation)
- Exercise: Standard care + 3-month exercise therapy
  Exercise: upper and lower extremity exercise
  Standard care: anticoagulation, compression, and ad-lib ambulation
Period: Overall Study
Arm/Group | Control | Exercise
Started (Randomized and completed baseline visit) | 48 | 54
Completed (Came in for 2-year follow-up visit) | 36 | 31
Not Completed | 12 | 23

BASELINE CHARACTERISTICS:
Population: Patients with acute DVT
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Exercise | Total
Number analyzed (Participants) | 48 | 54 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 52 (12) | 53 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 27 | 36 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 47 | 50 | 97
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 26 | 53
  White | 19 | 24 | 43
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 2 | 3
Villalta score [Mean (Standard Deviation); unit: units on a scale] — The Villalta score quantifies severity of symptoms and can be used to diagnose Post-Thrombotic Syndrome (PTS).
  Higher Villalta scores denote more severe symptoms and greater likelihood of PTS.
  The minimum possible score is 0, and the maximum possible score is 33. Population: Patients who underwent physical examination at baseline (some patients could not tolerate the physical examination necessary to ascertain Villalta score).
  units on a scale
    number analyzed (Participants) | 46 | 49 | 95
    (all) | 5.4 (4.5) | 4.2 (3.8) | 4.8 (4.1)
VEINES-QOL summary score [Mean (Standard Deviation); unit: units on a scale] — The VEINES-QOL summary score is calculated from the Venous Insufficiency Epidemiological and Economic Study (VEINES) Quality of Life (QOL) questionnaire, and it provides an estimate of the overall impact of deep venous thrombosis (DVT) on the patient's quality of life. A higher VEINES-QOL score indicates better quality of life.
  The minimum possible score is 25 and the maximum possible score is 117. Population: Patients who completed the VEINES-QOL questionnaire at baseline (some patients refused or were unable to complete the questionnaire).
  units on a scale
    number analyzed (Participants) | 42 | 49 | 91
    (all) | 84.2 (15.0) | 85.4 (16.8) | 84.8 (15.9)
SF-36 domain scores [Mean (Standard Deviation); unit: units on a scale] — The 36-Item Short Form survey (SF-36) produces 8 domain scores, each quantifying a different aspect of quality of life:
  * PF = Physical Functioning
  * RP = Role limitations due to Physical health problems
  * RE = Role limitations due to mental health or Emotional problems
  * VT = energy/fatigue/Vitality
  * MH = Mental Health/emotional well-being
  * SF = Social Functioning
  * BP = Bodily Pain
  * GH = General Health
  Higher scores denote better quality of life. For each domain score, the minimum possible score is 0 and the maximum possible score is 100. Population: Patients who completed the SF-36 questionnaire at baseline (some patients refused or were unable to complete the questionnaire).
  units on a scale
    PF domain score: number analyzed (Participants) | 43 | 49 | 92
    PF domain score | 44.9 (32.5) | 66.7 (29.7) | 56.5 (32.7)
    RP domain score: number analyzed (Participants) | 43 | 49 | 92
    RP domain score | 7.4 (10.2) | 9.8 (10.4) | 8.7 (10.3)
    RE domain score: number analyzed (Participants) | 43 | 49 | 92
    RE domain score | 15.1 (11.3) | 15.6 (10.7) | 15.6 (10.9)
    VT domain score: number analyzed (Participants) | 43 | 49 | 92
    VT domain score | 54.2 (27.9) | 59.9 (25.2) | 57.2 (26.5)
    MH domain score: number analyzed (Participants) | 43 | 49 | 92
    MH domain score | 68.4 (25.0) | 72.3 (20.3) | 70.5 (22.6)
    SF domain score: number analyzed (Participants) | 43 | 49 | 92
    SF domain score | 58.1 (35.7) | 65.6 (31.2) | 62.1 (33.4)
    BP domain score: number analyzed (Participants) | 43 | 49 | 92
    BP domain score | 47.9 (36.3) | 52.2 (29.4) | 50.2 (32.7)
    GH domain score: number analyzed (Participants) | 43 | 49 | 92
    GH domain score | 55.2 (25.3) | 62.5 (22.0) | 59.1 (23.8)
Thrombus volume [Mean (Standard Deviation); unit: mL] — Population: Patients for whom thrombus volume could be determined through imaging (thrombus volume could not be determined for some patients).
  mL
    number analyzed (Participants) | 42 | 47 | 89
    (all) | 3.0 (6.7) | 2.4 (4.4) | 2.7 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: 2-year Change in Villalta Score
Description: The Villalta score quantifies severity of symptoms and can be used to diagnose Post-Thrombotic Syndrome (PTS). The Villalta score quantifies severity of symptoms and can be used to diagnose Post-Thrombotic Syndrome (PTS). Higher Villalta scores denote more severe symptoms and greater likelihood of PTS.
  The outcome measure is not the score itself, but change in scores over time, calculated by subtracting the baseline score from the score at the 2-year follow-up.
  The range of the Villalta score is 0-33, so the minimum possible change is -33 and the maximum possible change is 33, with 0 indicating no change in Villalta scores (same score at baseline and at 2-year follow-up).
  An increase (positive change) in Villalta score indicates worsening symptoms, while a decrease (negative change) indicates improving symptoms.
Time Frame: Change from baseline to 2-year follow-up
Population: Patients who underwent physical examination at baseline and at the 2-year visit (some patients could not tolerate the physical examination necessary to ascertain Villalta score, and some patients did not complete a 2-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Exercise
Number analyzed (Participants) | 30 | 30
units on a scale | -1.5 (4.3) | -0.5 (3.7)
Statistical Analysis 1: Comparison: Control vs Exercise; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Net) = 1.0, 95% CI 2-sided [-1.1 to 3.1], Standard Error of Mean 1.0 — Mean difference = Exercise - Control

2. Primary Outcome: 2-year Change in VEINES-QOL Summary Score
Description: The VEINES-QOL summary score is calculated from the Venous Insufficiency Epidemiological and Economic Study (VEINES) Quality of Life (QOL) questionnaire, and it provides an estimate of the overall impact of deep venous thrombosis (DVT) on the patient's quality of life. A higher VEINES-QOL score indicates better quality of life.
  The outcome measure is not the score itself, but change in scores over time, calculated by subtracting the baseline score from the score at the 2-year visit.
  The range of the VEINES-QOL summary score is 25-117, so the minimum possible change is -92 and the maximum possible change is 92, with 0 indicating no change in VEINES-QOL scores (same score at baseline and at 2-year follow-up).
  An increase (positive change) in VEINES-QOL score indicates an improvement in quality of life, and a decrease (negative change) indicates worsening quality of life.
Time Frame: Change from baseline to 2-year follow-up
Population: Patients who completed the VEINES-QOL questionnaire at baseline and at the 2-year visit (some patients refused or were unable to complete the questionnaire, and some patients did not complete a 2-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Exercise
Number analyzed (Participants) | 23 | 30
units on a scale | 6.4 (8.2) | 6.9 (16.5)
Statistical Analysis 1: Comparison: Control vs Exercise; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [-7.1 to 8.0], Standard Error of Mean 3.5 — Mean difference = Exercise - Control

3. Secondary Outcome: 2-year Change in SF-36 Domain Scores
Description: The 36-Item Short Form survey (SF-36) produces 8 domain scores, each quantifying a different aspect of quality of life:
  * PF = Physical Functioning
  * RP = Role limitations due to Physical health problems
  * RE = Role limitations due to mental health or Emotional problems
  * VT = energy/fatigue/Vitality
  * MH = Mental Health/emotional well-being
  * SF = Social Functioning
  * BP = Bodily Pain
  * GH = General Health
  The outcome measure is not the score itself, but change in scores over time, calculated by subtracting the baseline score from the score at the 2-year visit.
  The range for each domain score is 0-100, so the minimum possible change is -100 and the maximum possible change is +100, with 0 indicating no change in domain scores (same score at baseline and at 2-year follow-up).
  An increase (positive change) in a domain score indicates improvement in that specific aspect of quality of life, and a decrease (negative change) indicates worsening quality of life in that domain.
Time Frame: Change from baseline to 2-year follow-up
Population: Patients who completed the SF-36 questionnaire at baseline and at the 2-year visit (some patients refused or were unable to complete the questionnaire, and some patients did not complete a 2-year follow-up visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Exercise
Number analyzed (Participants) | 24 | 30
units on a scale
  Change in PF domain score | 20.2 (30.9) | 14.4 (22.2)
  Change in RP domain score | 5.2 (13.8) | 10.2 (10.4)
  Change in RE domain score | 3.1 (11.5) | 5.8 (8.8)
  Change in VT domain score | 3.1 (26.9) | 8.7 (25.4)
  Change in MH domain score | 1.9 (22.4) | -0.7 (18.6)
  Change in SF domain score | 21.4 (28.4) | 17.5 (31.8)
  Change in BP domain score | 12.5 (34.8) | 22.0 (38.4)
  Change in GH domain score | 1.1 (22.0) | -2.4 (16.6)
Statistical Analysis 1: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Physical Functioning (PF) domain score; Test type: Superiority; p = 0.43, t-test, 2 sided; Mean Difference (Net) = -5.8, 95% CI 2-sided [-20.3 to 8.4], Standard Error of Mean 7.2 — Mean difference = Exercise - Control
Statistical Analysis 2: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Role limitations due to Physical health problems (RP) domain score; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Net) = 5.0, 95% CI 2-sided [-1.6 to 11.6], Standard Error of Mean 3.3 — Mean difference = Exercise - Control
Statistical Analysis 3: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Role limitations due to mental health or Emotional problems (RE) domain score; Test type: Superiority; p = 0.33, t-test, 2 sided; Mean Difference (Net) = 2.7, 95% CI 2-sided [-2.8 to 8.2], Standard Error of Mean 2.8 — Mean difference = Exercise - Control
Statistical Analysis 4: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the energy/fatigue/Vitality (VT) domain score; Test type: Superiority; p = 0.43, t-test, 2 sided; Mean Difference (Net) = 5.6, 95% CI 2-sided [-8.7 to 20.0], Standard Error of Mean 7.1 — Mean difference = Exercise - Control
Statistical Analysis 5: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Mental Health/emotional well-being (MH) domain score; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Net) = -2.6, 95% CI 2-sided [-13.8 to 8.6], Standard Error of Mean 5.6 — Mean difference = Exercise - Control
Statistical Analysis 6: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Social Functioning (SF) domain score; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Net) = -3.9, 95% CI 2-sided [-20.5 to 12.8], Standard Error of Mean 8.3 — Mean difference = Exercise - Control
Statistical Analysis 7: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the Bodily Pain (BP) domain score; Test type: Superiority; p = 0.35, t-test, 2 sided; Mean Difference (Net) = 9.5, 95% CI 2-sided [-10.7 to 29.7], Standard Error of Mean 10.1 — Mean difference = Exercise - Control
Statistical Analysis 8: Comparison: Control vs Exercise; Note that this analysis uses only 1 of the 8 SF-36 domain scores, the General Health (GH) domain score; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Net) = -3.5, 95% CI 2-sided [-14.1 to 7.0], Standard Error of Mean 5.3 — Mean difference = Exercise - Control

4. Secondary Outcome: 3-month Percent-change in Thrombus Volume
Description: Percent-change in thrombus volume (mL) is calculated by subtracting the baseline volume from the volume at the 3-month visit then dividing the result by the baseline volume and multiplying by 100.
  A negative change indicates a decrease in thrombus volume; i.e. the thrombus shrank in size and is therefore closer to complete resolution.
  A percent-change of -100% indicates complete thrombus resolution.
Time Frame: Change from baseline to 3-month follow-up
Population: Patients for whom thrombus volume could be determined through imaging at baseline and at the 3-month visit (thrombus volume could not be determined for some patients, and some patients did not complete a 3-month follow-up visit).
Measure: Mean (Standard Deviation); unit: Percent of baseline thrombus size
Arm/Group | Control | Exercise
Number analyzed (Participants) | 24 | 35
Percent of baseline thrombus size | -35.9 (138.1) | -69.8 (63.2)
Statistical Analysis 1: Comparison: Control vs Exercise; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Net) = -33.9, 95% CI 2-sided [-95.5 to 27.7], Standard Error of Mean 30.1 — Mean difference = Exercise - Control

5. Post Hoc Outcome: Villalta Score in People With vs Without Common Femoral Reflux
Description: Common femoral reflux (yes/no) is used as a measure of hemodynamics; determined through lower extremity Ultrasonography.
  The Villalta score quantifies severity of symptoms and can be used to diagnose Post-Thrombotic Syndrome (PTS). Higher Villalta scores denote more severe symptoms and greater likelihood of PTS. The minimum possible score is 0, and the maximum possible score is 33.
Time Frame: Baseline
Population: Patients who underwent physical examination (to ascertain Villalta score) as well as lower extremity Ultrasonography (to assess hemodynamics of the common femoral vein) at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Common Femoral Reflux: Patients with reflux in the common femoral vein.
- No Common Femoral Reflux: Patients without reflux in the common femoral vein.
Arm/Group | Common Femoral Reflux | No Common Femoral Reflux
Number analyzed (Participants) | 52 | 42
units on a scale
  Exercise: number analyzed (Participants) | 27 | 21
  Exercise | 3.9 (3.8) | 4.4 (3.9)
  Control: number analyzed (Participants) | 25 | 21
  Control | 4.1 (3.0) | 6.9 (5.5)
Statistical Analysis 1: Comparison: Common Femoral Reflux vs No Common Femoral Reflux; Test type: Superiority; p = 0.07, t-test, 2 sided; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.4 to 0.1], Standard Error of Mean 0.9 — Mean difference = Reflux - No reflux

6. Post Hoc Outcome: Time Required to Walk 400 Meters in Patients With vs Without PTS
Description: The 400-meter walk tests exercise capacity. Post-thrombotic syndrome (PTS) is defined as a Villalta score of 5 or higher.
Time Frame: Baseline
Population: Patients who underwent physical examination to ascertain Villalta score and completed 400-meter walk at baseline (some patients could not tolerate physical examination and some patients were unable to complete walk).
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- PTS (Villalta Score >=5): Post-thrombotic syndrome (Villalta score of 5 or higher)
- No PTS: No post-thrombotic syndrome (Villalta score between 0 and 4)
Arm/Group | PTS (Villalta Score >=5) | No PTS
Number analyzed (Participants) | 23 | 36
minutes
  Exercise: number analyzed (Participants) | 14 | 24
  Exercise | 5.9 (2.0) | 5.4 (1.1)
  Control: number analyzed (Participants) | 9 | 12
  Control | 4.9 (1.3) | 5.6 (1.4)
Statistical Analysis 1: Comparison: PTS (Villalta Score >=5) vs No PTS; Test type: Superiority; p = 0.91, t-test, 2 sided; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.8 to 0.9], Standard Error of Mean 0.4 — Mean difference = PTS - No PTS

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 years
Groups:
- Control: Standard care: anticoagulation, compression & ad-lib ambulation
  Control: Standard care: anticoagulation, compression & ad-lib ambulation
- Exercise: Standard care + Interventional Exercise therapy
  Exercise: Upper and Lower extremity exercise
  Standard care: anticoagulation, compression & ad-lib ambulation
Arm/Group | Control | Exercise
All-Cause Mortality (participants affected / at risk) | 6/48 | 3/54
Serious Adverse Events (participants affected / at risk) | 14/48 | 9/54
Other Adverse Events (participants affected / at risk) | 0/48 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=48) | Exercise (N=54)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1) — Chronic renal failure
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) — incarcerated ventral hernia
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) — Bowel obstruction by tumor
Colon Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Colon
Prostate Cancer (Renal and urinary disorders) | 1 (1) | 1 (1) — Prostate Cancer
Chronic Pain After Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Chronic pain after hip and ankle fracture
Cholecystectomy (Gastrointestinal disorders) | 0 (0) | 1 (1) — Gallbladder removal surgery
Neuroendocrine tumor (Endocrine disorders) | 0 (0) | 1 (1) — neuroendocrine tumor
Disseminated infection (Infections and infestations) | 1 (1) | 0 (0) — Disseminated infection with suspected Nocardia(bacteria)
Tumor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Lung Biopsy
Gun Shot Wound (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Gun Shot Wound
Respirtory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Pneumonia and Shortness of Breath
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pulmonary Embolism
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Upper Gastrointestinal Bleed
Intracranial bleeding (Vascular disorders) | 1 (1) | 0 (0) — Intracranial bleeding
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — worsening of bipolar disorder and homicidal ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT02148029/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT02148029/ICF_001.pdf